CLINICAL TRIAL: NCT03110679
Title: Randomized Double-blind Study on the Treatment of Osteoarthritis of the Bilateral Knee: Autologous Bone Marrow Concentrate vs. Hyaluronic Acid
Acronym: OA-bi-Blind
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OA-bi-Blind
Record Dates: First submitted 2017-03-30; First posted 2017-04-12 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-02

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; autologous bone marrow concentrate
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: autologous bone marrow concentrate vs. hyaluronic acid.
Who Masked: Participant, Investigator
Masking Description: cover the syringe to mask the contents
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- autologous bone marrow concentrate (Experimental): concentration of bone marrow taken from the patient's right tibia using Bio-MAC® suction catheter, company Biologic Therapies, Inc., and concentrated by centrifuge Bio.SPINTM Magellan®, company Biologic Therapies , Inc., and its injection in the intra-articular.
  Interventions: Biological: injection of autologous bone marrow concentrate
- hyaluronic acid. (Experimental): single injection of intra-articular hyaluronic acid 60mg (4 cc), and serve as a control.
  Interventions: Biological: injection of hyaluronic acid.

INTERVENTIONS:
Biological: injection of autologous bone marrow concentrate
  Arms: autologous bone marrow concentrate
Biological: injection of hyaluronic acid.
  Arms: hyaluronic acid.

SUMMARY:
OA-bi-Blind is a randomized double-blind study on the treatment of osteoarthritis of the Bilateral knee: autologous bone marrow concentrate vs. hyaluronic acid.

DETAILED DESCRIPTION:
a randomized, controlled, double-blind study and we will be evaluated and compared the clinical and radiological results of concentrated autologous bone marrow against the hyaluronic acid in patients with bilateral knee osteoarthrosis . In randomization, one knee will be treated with autologous bone marrow concentrate and other knee with hyaluronic acid, then every patient is considered both in control and treatment group, limiting the heterogenity between groups and will not be informed of the knee assigned to the treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, aged between 18 and 75 years;
2. Bilateral symptomatic knee osteoarthritis (Kellgren-Lawrence grade 1-4);
3. Failure after two months of conservative treatment;
4. Capacity and consent of patients to participate actively in the rehabilitation protocol, follow-up clinic and radiology protocol;
5. Signature of informed consent.

Exclusion Criteria:

1. Patients incapable of discernment;
2. Patients with malignancy
3. Patients with rheumatic diseases;
4. Patients with diabetes;
5. Patients with metabolic disorders of the thyroid;
6. Patients belonging abuse of alcohol, drugs or medications;
7. Patients with misalignment of the lower limbs than 10 °;
8. Body Mass Index> 40;
9. Patients with a history of trauma or intra-articular infiltration of therapeutic substances within 6 months prior to treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
International Knee Documentation Committee (IKDC)-Subjective score | Time Frame: 6 months
  Clinical improvement, measured by the change in scores IKDC Subjective

SECONDARY OUTCOMES:
International Knee Documentation Committee (IKDC)-Subjective score | Time Frame: 1,3,6, 12, 24 months evaluation
  Stability of the initial clinical improvement between 6 and 24 months
Knee Injury and Osteoarthritis Outcome Score (KOOS). | Time Frame: 1,3,6, 12, 24 months evaluation
  Stability of the initial clinical improvement between 6 and 24 months of the KOOS pain score

CONTACTS AND LOCATIONS:
Locations (1):
- Rizzoli Orthopaedic Institute, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No